CLINICAL TRIAL: NCT04358627
Title: Impact of Dexmedetomidine Infusion on the Time Course and Outcomes of Acute Respiratory Distress Syndrome (ARDS) in Patients Affected by the SARS-CoV-2 (COVID-19) Admitted to Critical Care Unit
Brief Title: Dexmedetomidine to Improve Outcomes of ARDS in Critical Care COVID-19 Patients
Acronym: COVID-DEX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: SPEC-M; SPEC-M COVID-19 (Other: Internal)
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Acute Respiratory Distress Syndrome; Inflammation; Dexmedetomidine; Cytokine Storm; Delirium, Emergence
MeSH Terms: conditions — Respiratory Distress Syndrome; Inflammation; Cytokine Release Syndrome; Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- DEXMEDETOMIDINE: Patients receiving dexmedetomidine continuous infusion since their admittance to ICU. Continuous checking of the primary and secondary outcomes
  Interventions: Drug: Dexmedetomidine Injectable Product
- No-DEXMEDETOMIDINE: Historical Control patients matched for ICU admittance diagnosis, age, and concomitant disease and medication state. No Dexmedetomidine. CONtinuous checking of primary outcomes

INTERVENTIONS:
Drug: Dexmedetomidine Injectable Product — continuous intravenous infusion of dexmedetomidine
  Other Names: DEX IV Sedation
  Groups: DEXMEDETOMIDINE

SUMMARY:
A continuous infusion of Dexmedetomidine (DEX) will be administered to 80 patients admitted to Critical Care because of signs of Respiratory Insufficiency requiring non-invasive ventilation. Measurements of respiratory performance and quantification of cellular and molecular inflammatory mediators. The primary outcome will be the avoidance of mechanical ventilation with secondary outcomes duration of mechanical ventilation, avoidance of delirium after sedation and association of mediators of inflammation to outcomes. Outcomes will be compared to a matched historical control (no DEX) series

DETAILED DESCRIPTION:
It will be an observational study, with no randomization. To evaluate the influence of Dexmedetomidine on the time course of ARDS in patients admitted to the ICU unit because of severe respiratory disease triggered by the SARS-CoV-2 (COVID-19) infection. Patients will be informed and asked to sign an Informed Consent Form.

Dexmedetomidine will be used as a sedative which is its admitted therapeutic indication in our country. Dosing will be according to its sedative properties as recommended by the manufacturer and regulation agencies. The only change is that we will study outcomes that have nothing to do with sedation but with a possible positive effect on the hyper-inflammatory state.

The study will be conducted in accordance with the "Orden SAS/3470/2009, of December 16, 2009. Government of Spain

Recruiting and Sample Size calculation We chose mortality as an endpoint to calculate sample size although our primary outcome is to minimize the requirements of mechanical ventilation. Mortality of patients admitted to the ICU because of SARS-CoV-2 (COVID-19) induced ARDS is 48%. Assuming a p value<0.05 and a power of 80%, to demonstrate a 10% decrease in mortality due to the effects of Dexmedetomidine 156 patients should be studied so there will two groups of 80 patients (cases vs historical controls).

However, due to the specific characteristics and the unknown duration of the pandemic, these numbers might not be definitive

Inclusion and Exclusion Criteria (see section)

Drug administrations Dexmedetomidine continuous intravenous infusion will be administered at 0.15 mcg/kg/h as a start and titrating according to sedative responses up to 1.5 mcg/kg/h (max admitted infusion rate)

Other sedatives (usually propofol and remifentanil) may be administered as per ICU protocol

Monitoring

* Ventilation parameters
* Invasive /non-invasive monitoring according to protocols
* The parasympathetic component of HRV will be estimated online by means of the Anesthesia Nociception Index (ANI, MDoloris Medical Systems, Lille, France).

Patient Management Patient management will be performed according to the clinical protocols of the Critical Care Units of Hospital CLINIC de Barcelona regarding the management of patients admitted to ICU because of the consequences of SARS-CoV-2 virus infection

Data Collection Demographic data including age, weight, gender, height, medical conditions, ICU severity score, SOFA score, medications, hemodynamic support, O2 fraction.

Besides regular protocolized monitoring measures for the purposes of the study it will be required:

* Routine Acid-Base equilibrium
* Routine hemogram
* Daily Citokine levels IL1b, IL6, TNFa, IL8, IL4, IL10
* Monocyte profiling Patient data will be kept anonymous except for the IP.

Outcomes to be measured are reported in their respective section

Data Analysis Analysis of the data collected includes the comparison of "primary and secondary outcomes data" acquired to a matched "historical control" with the same severity of ARDS from another COVID-19 + ICU patient with no administration of Dexmedetomidine. A "p" value less than 0.05 will be considered significant in the comparisons with the values of the "historical cohort".

Parametric or non-parametric statistical tests will be used to compare data from the control and study groups, depending on the distribution of such data.

Analysis of the time course of the mediators of inflammation sampled in the first 25 patients will be studied as changes from baseline. Mathematical models of the probability of each one or many of them to be associated with the outcomes of the study will be generated if possible

ELIGIBILITY:
Inclusion Criteria:

* Patients with respiratory insufficiency criteria candidates to non-invasive ventilation techniques (high flow oxygen masks, non-invasive mechanical ventilation)
* SpO2 (at FiO2: 0.21) ≤ 93% equivalent to SaO2/FiO2≤442
* PaO2/ FiO2 < 300
* Bilateral opacities consistent with pulmonary edema must be present and may be detected on CT or chest radiograph that must not be fully explained by cardiac failure or fluid overload, in the physician's best estimation using available information

Exclusion Criteria:

* Affected by autoimmune disease
* Under specific therapy with Monoclonal Antibodies targeting inflammatory mediators

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational study, with no randomization, to evaluate the influence of Dexmedetomidine on the time course of ARDS in patients admitted to the ICU unit because of severe respiratory disease triggered by the SARS-CoV-2 (COVID-19) infection.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation | expected within first three days (non conclusive due to lack of evidence yet)
  (Presence/Absence) requirement of mechanical ventilation

SECONDARY OUTCOMES:
Duration of mechanical ventilation | expected within first seven days (non conclusive due to lack of evidence yet)
  Duration of mechanical ventilation if it is required (hours from the start)
Delirium on recovery from sedation | First 24 hours after retiring dexmedetomidine sedation
  Delirium criteria as defined in DSM-4

IPD SHARING:
Plan to Share IPD: Undecided
We will share with interested researchers under the acceptance of our Ethics Committee